CLINICAL TRIAL: NCT05551273
Title: Safety, Tolerability, and Impact of Oral TLR8 Agonist Selgantolimod on HBsAg in Participants With Both Chronic Hepatitis B and HIV
Brief Title: Study of Oral TLR8 Agonist Selgantolimod on HBsAg in Participants With Both Chronic Hepatitis B and HIV
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A5394
Record Dates: First submitted 2022-09-09; First posted 2022-09-22 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Hepatitis B; HIV Infections
MeSH Terms: conditions — Hepatitis B; HIV Infections | interventions — selgantolimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Selgantolimod 3 mg once weekly for 24 weeks
  Interventions: Drug: Selgantolimod
- Arm B (Placebo Comparator): Matching Placebo for Selgantolimod once weekly for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Selgantolimod — 1.5 mg tablet
  Arms: Arm A
Drug: Placebo — Matching placebo tablet
  Arms: Arm B

SUMMARY:
The study aims to assess safety and tolerability of oral toll-like receptor (TLR) 8 agonist Selgantolimod (SLGN) administered for 24 weeks in participants with both CHB and HIV who have been receiving suppressive antiviral therapy for both viruses for ≥5 years and have qHBsAg level >1000 (3 log10) IU/mL at screening. The study will also evaluate if TLR8 stimulation with SLGN will reduce hepatitis B surface antigen (HBsAg) titers in the blood.

DETAILED DESCRIPTION:
A5394 is a phase II, double-blinded, placebo-controlled trial. Forty-eight study participants will be randomized 3:1 to receive SLGN or its placebo (36 active and 12 placebo), and randomization will be stratified by HBeAg status. One-half of the study participants will be HBeAg positive (n=24) at screening, and the other half will be HBeAg negative (n=24). All participants will remain on their non-study-provided antiviral therapy throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infection
2. Effective antiviral therapy for HIV (ART) and HBV that includes TDF, TAF, TDF/FTC, TDF/3TC (tenofovir disoproxil fumarate plus lamivudine), TAF/FTC, or entecavir (ETV), for ≥5 years immediately prior to study entry. ART is defined as including a minimum of two anti-HIV antivirals.
3. CD4+ cell count ≥350 cells/mm3
4. HIV-1 RNA <50 copies/mL measured on at least two occasions at least 12 weeks apart, with no documented value >200 copies/mL, over the 12 months prior to study entry.
5. Positive or negative HBeAg
6. Negative anti-HDV
7. Current CHB infection
8. HBV DNA level <50 IU/mL measured on at least two occasions at least 12 weeks apart, with no documented value ≥50 IU/mL, over the 12 months prior to study entry.
9. Quantitative HBsAg >1000 IU/mL
10. Hepatitis C virus (HCV) antibody negative, or if the participant is HCV antibody positive, an undetectable HCV RNA.
11. Participants age ≥18 years and ≤70 years at study entry
12. Participants must agree to stay on an effective antiviral therapy for HIV (ART) and HBV throughout the study.

Exclusion Criteria:

1. Receipt of treatment for HCV within 24 weeks prior to study entry
2. Evidence of advanced fibrosis or cirrhosis (Metavir ≥F3 or equivalent).
3. Current or prior history of clinical hepatic decompensation (e.g., ascites, encephalopathy, or variceal hemorrhage)
4. History of HCC or cholangiocarcinoma
5. Malignancy within 5 years prior to study entry. NOTE: A history of non-melanoma skin cancer (e.g., basal cell carcinoma or squamous cell skin cancer) is not exclusionary.
6. History of solid organ transplantation
7. Presence of any active or acute AIDS-defining opportunistic infections within 60 days prior to study entry
8. History of uveitis or posterior synechiae
9. Breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2025-10-29 (Actual); Study Completion 2026-04-29 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who experienced adverse events (AEs) | From study treatment initiation to Week 24
Proportion of participants who prematurely discontinued treatment due to adverse events (AEs) | From study treatment initiation to Week 24
Proportion of participants with ≥1 log10 IU/mL decline from baseline in quantitative HBsAg (qHBsAg) after SLGN treatment at Week 24 | At week 24

SECONDARY OUTCOMES:
Proportion of participants with ≥1 log10 IU/mL decline from baseline in qHBsAg at any time during the study after SLGN treatment Initiation | Baseline though week 48
Proportion of participants with ≥0.5 log10 IU/mL decline from baseline in qHBsAg after SLGN treatment at Week 24 | At week 24
Proportion of participants with ≥0.5 log10 IU/mL decline in qHBsAg from baseline at any time during the study after SLGN treatment initiation | Baseline though week 48
Proportion of participants who achieve HBsAg loss after SLGN initiation and who sustain HBsAg loss during follow-up | Baseline though week 48
Changes from baseline in qHBsAg levels at Weeks 4, 12, 24, 36, and 48 | At week 4, 12, 24, 36 and 48
Proportion of HBeAg positive participants at baseline who lose HBeAg at any time during the study | Baseline though week 48
Proportion of anti-HBe negative participants at baseline who develop anti-HBe at any time during the study | Baseline though week 48
Proportion of hepatitis B surface antibody (anti-HBs) negative participants at baseline who develop anti-HBs at any time during the study | Baseline though week 48
Detection of plasma HIV RNA >50 copies/mL at weeks 2, 4, 24, and 48 | At Weeks 2, 4, 24 and 48
Detection of serum HBV DNA >50 IU/mL at weeks 2, 4, 24, and 48 | At Weeks 2, 4, 24 and 48

CONTACTS AND LOCATIONS:
Locations (26):
- United States (16):
  - Alabama CRS, Birmingham, Alabama
  - UCSD Antiviral Research Center CRS, San Diego, California
  - The Ponce de Leon Center CRS, Atlanta, Georgia
  - Northwestern University CRS, Chicago, Illinois
  - Weill Cornell Chelsea CRS, New York, New York
  - Columbia P&S CRS, New York, New York
  - Weill Cornell Uptown CRS, New York, New York
  - Chapel Hill CRS, Chapel Hill, North Carolina
  - Greensboro CRS Site# 3203, Greensboro, North Carolina
  - Cincinnati Children's Hosp / Univ Hosp, Cincinnati, Ohio
  - Case CRS Site ID# 2501, Cleveland, Ohio
  - Ohio State University CRS, Columbus, Ohio
  - Univ of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt Therapeutics (VT) CRS, Nashville, Tennessee
  - Houston AIDS Research Team CRS, Houston, Texas
  - University of Washington AIDS CRS, Seattle, Washington
- Brazil (3):
  - Hospital Nossa Senhora da Conceicao CRS, Porto Alegre
  - Instituto de Pesquisa Clinica Evandro Chagas (IPEC) CRS Site ID# 12101, Rio de Janeiro
  - Instituto de Pesquisa Clinica Evandro Chagas (IPEC) CRS, Rio de Janeiro
- GHESKIO Institute of Infectious Diseases and Reproductive Health (GHESKIO - IMIS) CRS, Port-au-Prince, Haiti
- Barranco CRS, Lima, Peru
- De La Salle Health Science Institute Angelo King Medical Research Center (DLSHSI-AKMRC), Cavite, Philippines
- Soweto ACTG CRS, Johannesburg, Gauteng, South Africa
- Thailand (2):
  - Thai Red Cross AIDS Research Centre (TRC-ARC) CRS, Pathum Wan, Bangkok
  - Chiang Mai University HIV Treatment (CMU HIV Treatment) CRS, Chiang Mai
- Milton Park CRS, Milton Park, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the AIDS Clinical Trials Group by NIH
Access Criteria: With whom? Researchers who provide a methodologically sound proposal for use of the data that is approved by the AIDS Clinical Trials Group. For what types of analyses? To achieve aims in the proposal approved by the AIDS Clinical Trials Group. By what mechanism will data be made available? Researchers may submit a request for access to data using the AIDS Clinical Trials Group "Data Request" form at: https://actgnetwork.org/submit-a-proposal/. Researchers of approved proposals will need to sign an AIDS Clinical Trials Group Data Use Agreement before receiving the data